CLINICAL TRIAL: NCT06431373
Title: A Phase 3 Randomized, Double-Masked, Placebo-Controlled Study to Investigate the Safety and Efficacy of Oral Brepocitinib in Adults With Active, Non-Infectious Intermediate-, Posterior-, and Panuveitis
Brief Title: A Study of Brepocitinib in Adults With Active, Non-Infectious, Non-Anterior Uveitis
Acronym: CLARITY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Priovant Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PVT-2201-303
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Uveitis, Posterior; Uveitis, Intermediate; Uveitis
MeSH Terms: conditions — Uveitis, Posterior; Uveitis, Intermediate; Uveitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Brepocitinib PO QD
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo PO QD

INTERVENTIONS:
Drug: Brepocitinib PO QD — Brepocitinib PO QD
  Arms: Arm 1
Drug: Placebo PO QD — Placebo PO QD
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine the safety and efficacy of brepocitinib in participants with active, non-anterior (intermediate, posterior, or pan) non-infectious uveitis (NIU).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18-75 years old)
* Diagnosis of non-infectious uveitis (intermediate uveitis, posterior uveitis, or panuveitis)
* Active uveitic disease in at least 1 eye
* Weight > 40 kg with a body mass index ≤ 40 kg/m2

Exclusion Criteria:

Has confirmed or suspected current diagnosis of infectious uveitis History of or have:

1. Lymphoproliferative disorder
2. active malignancy
3. cancer within 5 years prior to screening (exceptions for basal cell carcinoma, squamous cell carcinoma, ductal carcinoma in situ of the breast, carcinoma in situ of the uterine cervix, or thyroid carcinoma.)
4. thrombosis or cerebrovascular ischemic event disease within the last 12 months
5. a high risk for herpes zoster reactivation
6. active or recent infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-09-11 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure on or after Period 1 Week 6 up to Period 1 Week 48 | 48 weeks

SECONDARY OUTCOMES:
Proportion of participants meeting treatment failure criteria on or after Period 1 Week 6 up to Period 1 Week 24 | 24 weeks
Change in logMAR BCVA in each eye from best state achieved at or prior to Period 1 Week 6 up to Period 1 Week 24 | 24 weeks
Change in central subfield thickness from best state achieved in each eye at or prior to Period 1 Week 6 up to Period 1 Week 24 | 24 weeks
Change in logMAR BCVA in each eye from best state achieved at or prior to Period 1 Week 6 up to Period 1 Week 48 | 48 Weeks
Change in central subfield thickness from best state achieved in each eye at or prior to Period 1 Week 6 up to Period 1 Week 48 | 48 weeks

CONTACTS AND LOCATIONS:
Locations (92):
- United States (47):
  - Clinical Trial Site, Phoenix, Arizona
  - Clinical Trial Site, Bakersfield, California
  - Clinical Trial Site, Beverly Hills, California
  - Clinical Trial Site, Fullerton, California
  - Clinical Trial Site, Irvine, California
  - Clinical Trial Site, La Jolla, California
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Modesto, California
  - Clinical Trial Site, Sacramento, California
  - Clinical Trial Site, Aurora, Colorado
  - Clinical Trial Site, Denver, Colorado
  - Clinical Trial Site, Fort Lauderdale, Florida
  - Clinical Trial Site, St. Petersburg, Florida
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Oak Park, Illinois
  - Clinical Trial Site, Carmel, Indiana
  - Clinical Trial Site, Prairie Village, Kansas
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Waltham, Massachusetts
  - Clinical Trial Site, Ann Arbor, Michigan
  - Clinical Trial Site, Detroit, Michigan
  - Clinical Trial Site, Minneapolis, Minnesota
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, Omaha, Nebraska
  - Clinical Trial Site, Palisades Park, New Jersey
  - NYU Langone Health, New York, New York
  - Clinical Trial Site, Rochester, New York
  - Clinical Trial Site, Durham, North Carolina
  - Clinical Trial Site, Winston-Salem, North Carolina
  - Clinical Trial Site, Cleveland, Ohio
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Portland, Oregon
  - Clinical Trial Site, Erie, Pennsylvania
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Greenville, South Carolina
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Austin, Texas
  - Clinical Trial Site, Bellaire, Texas
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Katy, Texas
  - Clinical Trial Site, Plano, Texas
  - Clinical Trial Site, Round Rock, Texas
  - Clinical Trial Site, San Antonio, Texas
  - Clinical Trial Site, Madison, Wisconsin
- Argentina (2):
  - Clinical Trial Site, Rosario, Santa Fe Province
  - Clinical Trial Site, Buenos Aires
- Australia (3):
  - Clinical Trial Site, Sydney, New South Wales
  - Clinical Trial Site, East Melbourne, Victoria
  - Clinical Trial Site, Nedlands, Western Australia
- Clinical Trial Site, Linz, Austria
- Clinical Trial Site, Leuven, VI-Brabant, Belgium
- Clinical Trial Site, Prague, Czechia
- Germany (6):
  - Clinical Trial Site, Mannheim, Baden-Wurttemberg
  - Clinical Trial Site, Bonn, North Rhine-Westphalia
  - Clinical Trial Site, Düsseldorf, North Rhine-Westphalia
  - Clinical Trial Site, Münster, North Rhine-Westphalia
  - Clinical Trial Site, Kiel
  - Clinical Trial Site, Mainz
- Clinical Trial Site, Thessaloniki, Greece
- Hungary (4):
  - Clinical Trial Site, Pécs, Baranya
  - Clinical Trial Site, Debrecen, Hajdú-Bihar
  - Clinical Trial Site, Budapest, Pest County
  - Clinical Trial Site, Budapest
- Israel (7):
  - Clinical Trial Site, Ashkelon
  - Clinical Trial Site, Haifa
  - Clinical Trial Site, Holon
  - Clinical Trial Site, Jerusalem
  - Clinical Trial Site, Kfar Saba
  - Clinical Trial Site, Poria – Neve Oved
  - Clinical Trial Site, Tel Aviv
- Italy (4):
  - Clinical Trial Site, Perugia, Umbria
  - Clinical Trial Site, Milan
  - Clinical Trial Site, Reggio Emilia
  - Clinical Trial Site, Roma
- Spain (4):
  - Clinical Trial Site, Barcelona, Catalonia
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Madrid
  - Clinical Trial Site, Valladolid
- United Kingdom (11):
  - Clinical Trial Site, London, England
  - Clinical Trial Site, Maidstone, Kent
  - Clinical Trial Site, Middlesbrough, North Yorkshire
  - Clinical Trial Site, Oxford, Oxfordshire
  - Clinical Trial Site, Sheffield, South Yorkshire
  - Clinical Trial Site, Birmingham, West Midlands
  - Clinical Trial Site, Bradford, Yorkshire
  - Clinical Trial Site, Birmingham
  - Clinical Trial Site, Bristol
  - Clinical Trial Site, Liverpool
  - Clinical Trial Site, Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://clarityuveitis.com/